CLINICAL TRIAL: NCT02978027
Title: Mentored Research on Improving Alcohol Brief Interventions in Medical Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: K23AA020865 (NIH); K23AA020865 (NIH)
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Alcohol Abuse
Keywords: motivational interviewing; brief alcohol intervention in primary care
MeSH Terms: conditions — Alcoholism | interventions — Crisis Intervention; Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brief Advice (Active Comparator): The brief advice protocol was designed by removing MI-consistent elements from the NIAAA Clinician's Guide. The protocol involves screening and assessment using the NIAAA pre-screen and single-question screen and assessing for quantity and frequency. Patients exceeding recommended limits receive feedback, information, and advice to cut down drinking to recommended levels. All patients are provided with a tip sheet on strategies for cutting down and encouraged to follow-up with a behavioral health provider with any questions or concerns.
  Interventions: Behavioral: Brief Advice
- NIAAA Clinician's Guide (Active Comparator): The NIAAA brief intervention was adapted directly from the NIAAA publication "Helping Patients Who Drink Too Much: A Clinician's Guide". The protocol screens using the NIAAA pre-screen and single-questions. Patients exceeding recommended limits receive feedback, information, and advice to cut down. For patients unwilling to make a change, the clinician restates their concern, encourages self reflection by asking the patient about reasons to cut down on drinking and barriers to change, and reaffirms willingness to help. For patients willing to make a change, the clinician helps the patient develop a plan to cut down within maximum limits, agree on specific steps and strategies, and provides a tip sheet on strategies for cutting down.
  Interventions: Behavioral: NIAAA Clinician's Guide
- Motivational Interviewing (MI) (Experimental): The MI intervention condition was also adapted from the NIAAA Clinician's Guide, with additional modification to include elements of MI. Clinicians normalize Screening and Brief Intervention (SBI) and ask the patient's permission before discussing alcohol use. The NIAAA pre-screen and single-question screen are administered. Assessment of quantity, frequency, and Alcohol Use Disorder symptoms is done using open questions. The ask-tell-ask technique is used to share feedback and exchange information regarding U.S adult drinking patterns. For patients low in readiness to make a change, clinicians build readiness using structured MI tools. For patients high in readiness to change, the ask-tell-ask technique is used to explore strategies for cutting down and develop an action plan.
  Interventions: Behavioral: Motivational Interviewing (MI)

INTERVENTIONS:
Behavioral: Brief Advice
  Arms: Brief Advice
Behavioral: NIAAA Clinician's Guide
  Arms: NIAAA Clinician's Guide
Behavioral: Motivational Interviewing (MI)
  Arms: Motivational Interviewing (MI)

SUMMARY:
The NIAAA estimates that 16% (40 million) of adults in the US are drinking at unsafe levels. More than 50% of alcohol health consequences occur in risky, non-dependent drinkers. Increasing the efficacy and efficiency of brief interventions in medical setting could significantly reduce the public health impacts of risky drinking. There is intense interest in conducting motivational interviewing (MI) informed brief interventions for risky alcohol use in medical settings, but little empirical information is available regarding which MI behavioral and interpersonal style components drive effectiveness. The field would benefit greatly from empirically-based Stage 1 treatment development and modeling studies to delineate the degree to which adding motivational interviewing components to brief intervention improves outcome.

DETAILED DESCRIPTION:
The NIAAA estimates that 16% (40 million) of adults in the US are drinking at unsafe levels, placing them at risk for a variety of physical, mental health, and social consequences. More than 50% of alcohol health consequences occur in risky, non-dependent drinkers. Increasing the efficacy and efficiency of brief interventions in medical setting could significantly reduce the public health impacts of risky drinking. Despite overall positive findings for brief interventions, there are high levels of variability in effects, with meta-analyses reporting significant unexplained heterogeneity in outcomes that is likely accounted for by differences in intervention components and strategies. There is intense interest in conducting motivational interviewing (MI) informed brief interventions for risky alcohol use in medical settings, but little empirical information is available regarding which MI behavioral and interpersonal style components drive effectiveness.

Following promising efficacy trials from counseling applications, MI was translated into brief (5-15 minute) interactions and subjected to randomized controlled trial methodology. Lack of mixed-methods, Stage 1 treatment development is evidenced by our inability to provide consistent delineation of key intervention components and mechanisms of action. Variability in these factors is likely responsible for the wide variability in effects observed in meta-analyses of brief interventions. Many MI skills and behaviors require significant training and supervision and increased patient-provider interaction time. The field would benefit greatly from empirically-based Stage 1 treatment development and modeling studies to delineate the degree to which adding motivational interviewing components to brief intervention improves outcome.

ELIGIBILITY:
Inclusion Criteria: patient in University of New Mexico Family and Community Medicine Clinic (e.g. Family Practice, Southeast Height, Northeast Height, University Clinic, South Valley), positive NIAAA single question screen (>0), AUDIT-C score <7, >18 years old, ability to read and speak English, and willing to be contacted for follow-up.

Exclusion Criteria: active suicidality, incarceration, obvious cognitive impairment, unable to provide informed consent, current involvement in an alcohol research study or people who are specifically seeking help for alcohol problems, and pregnancy or intent to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number days Exceeded Recommended Drinking Limits | 30 days

SECONDARY OUTCOMES:
Drinks Per Drinking Day | 30 days
Percent Days Abstinent | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hettema, PhD, Principal Investigator — The University of New Mexico Health Sciences Center
Locations (1):
- The University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hettema JE, Cockrell SA, Reeves A, Ingersoll KS, Lum PJ, Saitz R, Murray-Krezan CM, Carrejo VA. Development and differentiability of three brief interventions for risky alcohol use that include varying doses of motivational interviewing. Addict Sci Clin Pract. 2018 Feb 27;13(1):6. doi: 10.1186/s13722-017-0102-0. PMID 29482632